CLINICAL TRIAL: NCT05678452
Title: Comparative Study Between Safety and Efficacy of High Versus Low Power HOLEP in Enucleation of the Prostate; Prospective Randomized Double Blind Trial
Brief Title: Comparative Study Between Safety and Effectiveness of High Versus Low Power HOLEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: low and high power HOLEP
Record Dates: First submitted 2022-12-24; First posted 2023-01-10 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: HOLEP, Enucleation, Prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: HoLEP will be performed using 100W Versapulse, Luminis Inc., with 2J/25Hz for LP-HoLEP and 2J/50Hz for HP-HoLEP.
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LP-HoLEP (Active Comparator): 2J/25Hz setting
  Interventions: Procedure: HOLEP for treating BPH
- HP-HoLEP. (Active Comparator): 2J/50Hz setting
  Interventions: Procedure: HOLEP for treating BPH

INTERVENTIONS:
Procedure: HOLEP for treating BPH — HoLEP will be performed using 100W Versapulse, Luminis Inc., with 2J/25Hz for LP-HoLEP and 2J/50Hz for HP-HoLEP.

SUMMARY:
Holmium laser enucleation (HOLEP) has became a standard of treatment of large prostates that indicates surgery. HOLEP is widely used nowadays. Many settings are used but no optimal setting was world wide adopted. The aim of this trial is to assess the Low-power Holmium laser enucleation of the prostate (LP-HoLEP)and compare to high-power (HP-HoLEP) for enucleation efficiency pertaining to the advantages of lower cost and minimal postoperative dysuria, storage symptoms, and negative sexual impact.

ELIGIBILITY:
Inclusion Criteria:

* large prostate indicated for surgical intervention.

Exclusion Criteria:

* prostate cancer
* recurrent adenomas
* associated neurologic factors that may affect outcomes (e.g., neurogenic bladder)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Enucleation Efficiency | 3 hours
  Enucleated weight/min will be evaluated.

SECONDARY OUTCOMES:
Dysuria will be assessed by dysuria visual analog scale | 2 weeks
  burning micturation after the procedure. Dysuria will be assessed by dysuria visual analog scale
The complications of both techniques | 3 months
  The complications will be classified according to the modified Clavien classification system.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided